CLINICAL TRIAL: NCT04079634
Title: Esophageal Temperature Management During Cryo AF Ablation
Brief Title: Esophageal Temperature Management During Cryo AF Ablation (EnsoETM)
Acronym: EnsoETM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Attune Medical (Other)
Responsible Party: Principal Investigator, Nishant Verma, Assistant Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00209610
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will not be informed if they were randomized to control or treatment until Month 2 follow-up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Placement of study device (EnsoETM) for temperature management
  Interventions: Device: Esophageal warming
- Control (Active Comparator): Placement of standard temperature probe
  Interventions: Device: Control

INTERVENTIONS:
Device: Esophageal warming — Use of EnsoETM for esophageal warming to limit injury during atrial fibrillation ablation procedure
  Arms: Treatment
Device: Control — Standard temperature probe monitoring
  Arms: Control

SUMMARY:
The purpose of this pilot study is to determine if esophageal warming using the Attune Medical Esophageal Heat Transfer Device (EnsoETM) limits the frequency or severity of thermal injury during cryoballoon ablation of atrial fibrillation.

DETAILED DESCRIPTION:
Catheter ablation of atrial fibrillation (AF) has become a common ablation procedure performed worldwide. The cornerstone of this procedure is pulmonary vein isolation (PVI). PVI can be achieved by multiple methods, the two most common being radiofrequency (RF) and cryoablation. Energy delivery may extend beyond the atrial myocardium and result in damage to adjacent structures, including the esophagus. Atrio-esophageal fistula (AEF) is a rare, but a well-recognized complication of percutaneous AF ablation. The occurrence rate of esophageal injury has varied depending on the reporting center, timing of endoscopy, and the ablation technique utilized. Esophageal ulceration is likely the initial injury that leads to AEF formation and is probably present within hours to days of the ablation procedure.

The Attune Medical Esophageal Heat Transfer Device (EnsoETM) is a non-sterile, multi-lumen silicone tube placed in the esophagus for the purpose of cooling or warming a patient while simultaneously allowing gastric decompression and drainage. For this study, the EnsoETM tube will be used during cardiac ablation procedures for the intended indication of patient temperature management using approved settings/parameters as detailed in the product instructions for use document. EnsoETM is an FDA approved device.

This prospective, randomized study will include 40 patients with symptomatic AF undergoing index PVI under general anesthesia at Northwestern Memorial Hospital. Patients will be randomized in a 1:1 fashion with 20 patients (Group A) randomized to undergo the ablation procedure with esophageal warming and the other 20 patients (Group B) will serve as the control group and will not have the EnsoETM device used. All patients will undergo esophagogastroduodenoscopy (EGD) 1-2 days following the ablation procedure to evaluate for esophageal injury.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above the age of 18 years old.
2. Patients with the diagnosis of atrial fibrillation undergoing clinically indicated de-novo AF ablation procedure.
3. Patients must be willing to provide informed consent.

Exclusion Criteria:

1. Patients with contraindication to EGD.
2. History of prior AF ablation procedures.
3. Significant co-morbidities that preclude standard ablation procedure.
4. Patient is ineligible for EnsoETM placement due to:

   * Known esophageal deformity or evidence of esophageal trauma (for example history of esophagectomy, previous swallowing disorders, achalasia).
   * Known ingestion of acidic or caustic poisons within the prior 24 hours.
   * Patients with <40 kg of body mass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nishant Verma, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF
Time Frame: Within one year of enrollment closure
Access Criteria: Consent will be posted to ClinicalTrials.Gov

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 23 | 19
Completed | 23 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 7 | 19
  >=65 years | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (11.0) | 66.6 (8.4) | 65.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 14 | 16 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23 | 19 | 42
Hypertension (HTN) [Number; unit: participants] | 12 | 13 | 25
Diabetes [Number; unit: participants] | 2 | 1 | 3
Coronary Artery Disease (CAD) [Number; unit: participants] | 2 | 1 | 3
Cerebrovascular Accident (CVA) [Number; unit: participants] | 3 | 2 | 5
Paroxysmal Atrial Fibrillation (AF) [Number; unit: participants] | 14 | 11 | 25
Persistent Atrial Fibrillation (AF) [Number; unit: participants] | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Esophageal Thermal Injury
Description: Endoscopic evidence of thermal injury
Time Frame: Post-Procedure Day 1
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 23 | 19
participants | 8 | 1
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Other; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Description: Information on all adverse events will be recorded immediately in the source document, and also in the appropriate adverse event case report form (CRF). All clearly related signs, symptoms, and clinically significant abnormal diagnostic procedures results should be recorded in the source document. All adverse events occurring during the study period (consent through 3 month follow up) will be recorded.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 0/23 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT04079634/Prot_SAP_002.pdf
  • Informed Consent Form (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT04079634/ICF_001.pdf